CLINICAL TRIAL: NCT00477191
Title: Effects of TNF-alpha Antagonism (Etanercept) in Patients With the Metabolic Syndrome and Psoriasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruitment.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Alexandra Kimball, Director, Clinical Unit for Research Trials in Skin, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-P-000494
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Psoriasis; Metabolic Syndrome; Hyperlipidemia; Obesity; Hypertension
Keywords: psoriasis; metabolic syndrome; Syndrome X; diabetes; insulin resistance; obesity; hypertension; hyperlipidemia; hypercholesterolemia
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome; Hyperlipidemias; Obesity; Hypertension; Microvascular Angina; Diabetes Mellitus; Insulin Resistance; Hypercholesterolemia | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental): Etanercept
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — TNF-alpha antagonist 50 mg twice a week x 3 mos and the 50 mg once a week for 3 months.
  Other Names: Enbrel

SUMMARY:
People with psoriasis have significantly higher rates of obesity, diabetes, heart failure and high blood pressure than the general public. The purpose of this study is to determine how substances produced in the fat (inflammatory markers) relate to the risk of heart disease in people with the metabolic syndrome and psoriasis. People with metabolic syndrome have insulin resistance, increased waist size, high blood pressure, or high cholesterol.

DETAILED DESCRIPTION:
People with psoriasis have significantly higher rates of obesity, diabetes, heart failure and high blood pressure than the general public. The purpose of this study is to determine how substances produced in the fat (inflammatory markers) relate to the risk of heart disease in people with the metabolic syndrome and psoriasis. People with metabolic syndrome have insulin resistance, increased waist size, high blood pressure, or high cholesterol. Insulin resistance means that the body does not respond well to the insulin in your blood. Therefore, both blood levels of insulin and glucose (sugar) are high.

This causes inflammation (irritation) in the body. Inflammation can cause an unhealthy response in your body and blood vessels, and can lead to blockages in the heart and other vessels.

TNF-alpha is a substance made by fat and inflammatory cells that helps cause inflammatory reactions. TNF-alpha is thought to be important in causing psoriasis. The drug Etanercept blocks TNF-alpha's actions, and has been approved by the Food and Drug Administration (FDA) for the treatment of psoriasis. We think that Etanercept may also reduce the inflammation associated with metabolic syndrome and decrease the risk of heart disease. All subjects in this study will receive etanercept.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Subject willing and able to give informed consent.
3. Adult patients with chronic moderate to severe plaque psoriasis who are candidates for systemic therapy or phototherapy.
4. PASI > 10 and BSA affected with psoriasis > 10.
5. Abdominal obesity defined by waist hip ratio > 0.90 for men and > 0.85 for women and BMI ³ 30 kg/m2

Exclusion Criteria:

* On insulin or other diabetes (anti-hyperglycemic) medication
* Congestive Heart Failure
* Heart Attack, Stroke or Transient Ischemic Attack in last 3 months
* Unstable angina
* Pulmonary disease requiring oxygen
* SLE, optic neuritis, transverse myelitis, epilepsy
* Positive PPD
* Scheduled for upcoming surgery
* Known immunosuppression (for example, HIV)
* Known autoimmune disease
* Hepatitis B or Hepatitis C
* Pregnant or nursing
* Renal insufficiency (Creatinine >1.5)
* Latex allergy
* Use of live vaccination in past 90 days
* Organ transplantation
* History of severe infection
* History of malignancy (except cured non-melanoma skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra B Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital, Brigham & Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Etanercept
Started | 18
Completed | 13
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Psoriasis patients with MetS
Groups:
- Etanercept: Etanercept
  Etanercept: TNF-alpha antagonist 50 mg twice a week x 3 mos and then 50 mg once a week for 3 months.
Arm/Group | Etanercept
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 38.9 (5.6)
Psoriasis Area Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — The PASI is a measure of psoriatic disease severity taking into account qualitative lesion characteristics (erythema, thickness, and scaling) and degree of skin surface area involvement on defined anatomical regions. PASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement).
  units on a scale | 16.9 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in CRP Levels From Baseline to 6 Months of Treatment in Subjects With Psoriasis and Metabolic Syndrome
Description: Analyzing the difference in C reactive protein levels from baseline to month 6 in subjects with Psoriasis and Metabolic Syndrome
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Etanercept
Number analyzed (Participants) | 13
ng/mL | 5.3 (4.2)

2. Secondary Outcome: Change in Plasma Glucose in Subjects With Psoriasis and Metabolic Syndrome
Description: Analyzing the difference in plasma glucose in subjects with Psoriasis and Metabolic Syndrome between baseline and month 6.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Etanercept
Number analyzed (Participants) | 13
mg/dl | 13 (56)

3. Secondary Outcome: Change of Endothelial Function by Measurement of Flow-mediated Vasodilation Using the Reactive Hyperemia Index (RHI) in 6 Months
Description: Reactive hyperemia index (RHI) is a measure of endothelial dysfunction using noninvasive peripheral arterial tonometry (PAT). It is a ratio of the post-to-pre occlusion PAT amplitude of the tested arm, divided by the post -to-pre occlusion ratio of the control arm. RHI less than 1.67 is considered sign of endothelial dysfunction. The possible range of scores is 1 to 3 and a lower score has a worse outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 13
units on a scale | 1.57 (0.21)

4. Secondary Outcome: Change in the Safety and Tolerability of Etanercept in Patients With Psoriasis and Metabolic Syndrome Over a 6-month Period.
Description: Analyzing the safety and tolerability of Etanercept which is being measured through the number of adverse events related to Entanercept over a 6-month period.
Time Frame: 6 months
Measure: Number; unit: number of events
Arm/Group | Etanercept
Number analyzed (Participants) | 13
number of events | 6

ADVERSE EVENTS:
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etanercept (N=13)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Viral Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
It was likely underpowered to detect small changes in laboratory and exam measures. Patients were only evaluated after a 6 month course of etanercept therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No